CLINICAL TRIAL: NCT00612092
Title: Prospective Randomized Trial On RadiaTion Dose Estimates Of CT AngIOgraphy In PatieNts Scanned With A Sequential Scan Protocol
Acronym: PROTECTION-III
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Deutsches Herzzentrum Muenchen (Other)
Responsible Party: PD Dr. Joerg Hausleiter, Deutsches Herzzentrum
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: GE IDE No. R00308
Record Dates: First submitted 2008-01-28; First posted 2008-02-11 (Estimated); Last update posted 2008-08-27 (Estimated); Status verified 2008-08

CONDITIONS: Coronary Disease
Keywords: Coronary CT angiography; Radiation dose estimates
MeSH Terms: conditions — Coronary Disease

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Standard spiral CT protocol
  Interventions: Radiation: Spiral image acquisition
- 2 (Active Comparator): Sequential CT protocol
  Interventions: Radiation: sequential image acquisition

INTERVENTIONS:
Radiation: Spiral image acquisition — standard spiral scan protocol
  Arms: 1
Radiation: sequential image acquisition — sequential CT scan protocol
  Arms: 2

SUMMARY:
The objective of this study is to compare radiation dose of a standard spiral scan with the a new sequential scan protocol. We hypothesize that the sequential scan protocol is associated with a reduction in dose estimates of at least 20%, while the diagnostic image quality is not inferior.

Secondary endpoints of the study include quantitative image quality parameters, diagnostic accuracy for spiral versus sequential studies compared to invasive angiography in patients who underwent subsequent invasive coronary angiography.

DETAILED DESCRIPTION:
All patients scheduled for a coronary CT scan are screened for inclusion and exclusion criteria. Patients are included if they have stable sinus rhythm (heart rate <75 bpm for dual source CT and <65 bpm for 64-slice CT). Informed signed consent is obtained from these patients and the CT scan is prepared. After topogram scan and the native scan for Ca-Scoring, patients are randomized in two groups with the use of sealed envelopes. After that contrast-enhanced coronary CT angiography is performed with the standard spiral protocol or with the sequential protocol.

The CT examination is evaluated by two experienced investigators on a per-vessel basis and all results and study-related data are collected in a dedicated database. For assessment of image quality, a previously established 4-point score system is used and quantitative image quality parameters are measured.

A 30 day follow-up after the CT examination aims to evaluate if patients underwent invasive coronary angiography or were scheduled for a myocardial stress / perfusion test (such as stress-echocardiography, myocardial scintigraphy or stress perfusion imaging by MRI).

ELIGIBILITY:
Inclusion Criteria:

* patients with an indication for a coronary CT angiography (planned evaluation of the coronary arteries)
* stable sinus rhythm
* heart rate < 75 bpm with dual-source CT or < 65 bpm with single-source CT
* signed informed consent

Exclusion Criteria:

* non-ECG triggered studies
* non-coronary CTA studies, e.g. bypass graft CTAs, pre- or post EP studies, CABG planning studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2008-05; Primary Completion 2009-01 (Estimated); Study Completion 2009-02 (Estimated)

PRIMARY OUTCOMES:
Compared with a helical scan protocol the use of a sequential scan protocol is associated with a comparable diagnostic image quality, while the radiation dose estimates are significantly reduced. | 1 month

SECONDARY OUTCOMES:
impact of the sequential scan protocol on quantitative image quality parameters, e.g. image noise, signal and contrast intensity, signal- and contrast-to-noise-ratios | 30 days
diagnostic accuracy (sensitivity, specificity as well as positive and negative predictive values) for studies scanned with helical vs. sequential scan protocol when compared with invasive coronary angiography on a per-vessel based analysis | 30 days
frequency of non-diagnostic CTA studies when comparing studies scanned with the helical vs. the sequential scan protocol | 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Joerg Hausleiter, MD, Principal Investigator — Deutsches Herzzentrum Muenchen
Locations (1):
- Deutsches Herzzentrum Muenchen, Munich, Germany

REFERENCES:
- [Derived] Hausleiter J, Meyer TS, Martuscelli E, Spagnolo P, Yamamoto H, Carrascosa P, Anger T, Lehmkuhl L, Alkadhi H, Martinoff S, Hadamitzky M, Hein F, Bischoff B, Kuse M, Schomig A, Achenbach S. Image quality and radiation exposure with prospectively ECG-triggered axial scanning for coronary CT angiography: the multicenter, multivendor, randomized PROTECTION-III study. JACC Cardiovasc Imaging. 2012 May;5(5):484-93. doi: 10.1016/j.jcmg.2011.12.017. PMID 22595156